CLINICAL TRIAL: NCT04866901
Title: Examining the Interactive Effects of Mindfulness and Slow-paced Breathing on Stress Physiology: A Pilot Study
Brief Title: Interactive Effects of Mindfulness and Slow-paced Breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Michael R. Goldstein, Research Fellow, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020P000992
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Stress; Stress, Psychological; Stress Physiology; Sleep; Slow Breathing
Keywords: stress; slow-paced breathing; breath training; mindfulness; yogic breathing; wellness; stress-management
MeSH Terms: conditions — Stress, Psychological; Hypoventilation | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Slow-Paced Breathing (SPB) (Experimental): Participants will first be provided with a brief overview of the science of breathing and benefits for autonomic regulation. Then, participants will receive specific practice instruction and guided breathing at a rhythm of 6 breaths/min (4-6 count) via auditory tones. Each participant will be encouraged to breathe as comfortably and effortlessly as possible, while keeping the lungs moving in accordance with the audio guidance. The accompanying training and daily instruction reminder will emphasize the importance of following the specific rhythm of breathing, without regard to thoughts or inner experience. A soft but firm tone of voice will be employed to minimize likelihood of relaxing effects, while maintaining similarity to the tone of voice used in the other conditions.
  Interventions: Behavioral: Slow-Paced Breathing (SPB)
- Mindfulness (M) (Experimental): Procedures are based on Berghoff et al., providing a brief history of mindfulness practices, definitions, instructions for practice, common challenges, and recommendations. An audio recording will then guide the mindfulness practice. Specific to this study, in order to further distinguish the three conditions, the guided audio recording will emphasize the importance of attending to the quality of experience while not changing or attending to breathing patterns.
  Interventions: Behavioral: Mindfulness (M)
- Yogic Breathing (SPB+M) (Experimental): Information from the other two conditions will be synthesized with the aim of eliciting attention to the same breathing instruction used for SPB, while also observing the quality of experience during the practice, as conducted for M.
  Interventions: Behavioral: Yogic Breathing (SPB+M)

INTERVENTIONS:
Behavioral: Slow-Paced Breathing (SPB) — see arm description
  Arms: Slow-Paced Breathing (SPB)
Behavioral: Mindfulness (M) — see arm description
  Arms: Mindfulness (M)
Behavioral: Yogic Breathing (SPB+M) — see arm description
  Arms: Yogic Breathing (SPB+M)

SUMMARY:
The purpose of this study is to better understand specific stress-management practices on mood, sleep, and physiology. Participants will be assigned to one of three interventions (they all active interventions - none are a "wait-list"). Each intervention asks participants to engage in a daily practice of 20 minutes per day for 8 weeks. Questionnaires and measures of heart rate and blood pressure will be collected at the start and end of the 8 weeks, including a virtual laboratory visit.

DETAILED DESCRIPTION:
Slow-paced breathing (SPB), mindfulness (M), and their combination (SPB+M) in the form of yoga, yogic breathing, Tai Chi, Qigong, and other practices are considered distinct forms of intervention, yet are often considered inextricably linked and overlapping in their effects on the autonomic nervous system. Although the scientific community continues to build understanding of autonomic mechanisms that might be unique to SPB, M, and their interaction (SPB+M), no studies we are aware of have attempted to directly compare these three forms of intervention in a controlled fashion that enables a 'dismantling' framework of interpretation.

The goal of this pilot project is to compare the separate and combined effects of SPB and M on autonomic function. We will test the feasibility of a three-arm intervention trial (N=5 per group), involving 20-min daily practice for 8 weeks, with multimodal ambulatory autonomic measurement before and after intervention. We will first focus on a healthy young adult population to then inform translation to hypertension, insomnia, and other clinical groups.

Aim 1: Distinguish SPB, M, and SPB+M training in terms of breathing rate and subjective mindfulness.

Aim 2: Obtain pilot data comparing the three interventions in terms of autonomic regulation using both conventional metrics and non-linear dynamics.

Aim 3: Develop methods to examine relationships across domains of autonomic regulation, stress, and sleep for the three interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-24 years.

Exclusion Criteria:

* Active infection/disease
* Current untreated mental or physical health condition deemed likely to interfere with ability to complete study procedures (determined by study staff consensus)
* Current use of medications with known effects on stress physiology (antidepressants [SSRI, SNSI, NDRI, atypical, TCA, MAOI], anitpsychotics, benzodiazepines, non-benzodiazepine receptor agonists, melatonin and melatonin receptor agonists, orexin/hypocretin receptor antagonists, barbiturates, mood stabilizers, anticonvulsants, anticholinergics, first generation antihistamines, and stimulants including NRI, antihypertensives, opioids, or systemic corticosteroids)
* Moderate/substantial prior meditation, yoga, or other mind-body practice self-reported as a self-rating of 5 or higher on a scale of 0-10 asking "How experienced are you with meditation, yoga, or other mind-body interventions?"

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Breathing rate | 8-weeks (post-intervention), 15 minute practice session during the virtual laboratory visit
  Participants will wear a Polar H10 chest strap heart rate monitor during training and daily practice, and breathing rate will be derived from the HR interbeat interval series. We expect participants randomized to SPB and SPB+M to show slower breathing rates compared to M during a recorded practice session at 8-weeks.
Five Facet Mindfulness Questionnaire (FFMQ) | 8-weeks (post-intervention) completed electronically prior to virtual laboratory visit
  We expect M and SPB+M to more highly report qualities of experience consistent with mindfulness. Primary outcome will focus on total score, summing across the five facets (total score range: 39-195; higher scores reflect higher mindfulness ratings).

SECONDARY OUTCOMES:
Systolic blood pressure | 8-weeks (post-intervention), stress induction task (Stroop test) during the virtual laboratory visit
  We hypothesize that the combined SPB+M condition will show a pattern of lower systolic BP.
Heart rate variability (normalized high-frequency power, HFnu) | 8-weeks (post-intervention), stress induction task (Stroop test) during the virtual laboratory visit
  We hypothesize that the combined SPB+M condition will show a pattern of higher HFnu.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Goldstein, PhD, Principal Investigator — Beth Israel Deaconess Medical Center, Harvard Medical School
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No